CLINICAL TRIAL: NCT02948777
Title: Effects of PCSK9 Inhibition by Evolocumab on Postprandial Lipid Metabolism in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marja-Riitta Taskinen (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor-Investigator, Marja-Riitta Taskinen, Professor, emerita, Clinical Research Institute HUCH Ltd
Organization: Clinical Research Institute HUCH Ltd (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVOLKIN
Record Dates: First submitted 2016-10-27; First posted 2016-10-28 (Estimated); Results first posted 2021-10-11 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: apolipoprotein, CVD, chylomicrons, evolocumab, kinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Evolocumab (Experimental): Evolocumab 140 mg subcutaneous injection once every 2 weeks for 12 weeks
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab
  Other Names: Repatha

SUMMARY:
Postprandial lipemia is highly prevalent in type 2 diabetes subjects even with normal fasting triglyceride values. Humans are mostly in a postprandial rather than in a fasting state and therefore non-fasting triglyceride values reflect more accurately the continuous exposure of arterial wall to the substantial cholesterol load from remnant particles. Evolocumab lowers blood LDL-cholesterol. This study evaluates the effect of evolocumab on postprandial lipid metabolism in type 2 diabetes. All participants in this study receive evolocumab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (non-fertile or using a medically approved birth control method) overweight/obese subjects with Type 2 Diabetes Mellitus treated with lifestyle counselling and a stable metformin dose for at least three months
* age 18-77 yrs.
* body mass index 25-40 kg/m2
* triglycerides between 1.5-4.5 mmol/L and low-density-lipoprotein cholesterol >1.8 but ≤4.0 mmol/L (on Atorvastatin 20 mg/day)
* glycohemoglobin: ≤9%.
* Each patient will attend a pre-screening visit (at week -5) where eligibility criteria will be evaluated. If the patient uses another statin than atorvastatin (20 mg) at screening visit the used statin is stopped and atorvastatin 20 mg will be initiated. If the patient is not using any statin, atorvastatin 20 mg will be initiated and the lipid values will be checked after 4 weeks when all inclusion/exclusion criteria will be assessed.

Exclusion Criteria:

* Type 1 diabetes
* apolipoprotein E2/2 phenotype
* alanine transaminase / aspartate transaminase > 3× upper limit of normal
* creatinine kinase>3× upper limit of normal
* glomerular filtration rate <60 ml/min
* clinically significant thyroid-stimulating hormone outside the normal range
* body mass index >40 kg/m2
* glycohemoglobin > 9.0 %
* fasting triglycerides > 4.5 mmol/l
* total cholesterol > 7.0 mmol/l
* positive urine or serum pregnancy test
* untreated or inadequately treated hypertension defined as blood pressure >160 mmHg systolic and/or >105 mmHg diastolic, use of thiazide diuretics at a dose of ≥25 mg/day
* subject not on a stable dose of atorvastatin (20 mg/ day before randomization)
* lipid-lowering drugs other than statins within 3 months
* any other diabetes medication except diet + metformin
* history/diagnosis of diabetes nephropathy / retinopathy
* current smoking
* weekly alcohol use over 24 doses for men and 16 for women
* history of myocardial infarction, acute coronary syndrome or coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting) within the last 6 mos.
* planned revascularization (eg coronary artery bypass grafting, percutaneous coronary intervention, carotid or peripheral revascularization procedures) within 3 months of screening
* New York Heart Association class III/IV congestive heart failure persisting despite treatment
* history of hemorrhagic stroke
* hypersensitivity to (evolocumab or) any of the excipients found in the drug product
* use of estrogen therapy
* current use of antithrombotic or anticoagulant therapy
* known bleeding tendency that would be an contraindication to heparin test
* history of cancer within the past 5 years (except for adequately treated basal cell skin cancer, squamous cell skin cancer or in situ cervical cancer)
* women of childbearing potential not protected by effective birth control method and/or not willing to be tested for pregnancy
* patient considered by the investigator or any sub-investigator as inappropriate for this study for any reason

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-10; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marja-Riitta Taskinen, Prof., PI, Principal Investigator — Clinical Research institute Huch, Ltd and University of Helsinki; Jan Boren, Prof., co-PI, Principal Investigator — University of Gothenburg and Sahlgrenska University Hospital
Locations (1):
- Helsinki University Hospital, Biomedicum 2U, Helsinki, Finland

REFERENCES:
- [Result] Taskinen MR, Bjornson E, Kahri J, Soderlund S, Matikainen N, Porthan K, Ainola M, Hakkarainen A, Lundbom N, Fermanelli V, Fuchs J, Thorsell A, Kronenberg F, Andersson L, Adiels M, Packard CJ, Boren J. Effects of Evolocumab on the Postprandial Kinetics of Apo (Apolipoprotein) B100- and B48-Containing Lipoproteins in Subjects With Type 2 Diabetes. Arterioscler Thromb Vasc Biol. 2021 Feb;41(2):962-975. doi: 10.1161/ATVBAHA.120.315446. Epub 2020 Dec 24. PMID 33356392
- [Result] Taskinen MR, Bjornson E, Andersson L, Kahri J, Porthan K, Matikainen N, Soderlund S, Pietilainen K, Hakkarainen A, Lundbom N, Nilsson R, Stahlman M, Adiels M, Parini P, Packard C, Boren J. Impact of proprotein convertase subtilisin/kexin type 9 inhibition with evolocumab on the postprandial responses of triglyceride-rich lipoproteins in type II diabetic subjects. J Clin Lipidol. 2020 Jan-Feb;14(1):77-87. doi: 10.1016/j.jacl.2019.12.003. Epub 2019 Dec 12. PMID 31917184
- [Result] Zech LA, Grundy SM, Steinberg D, Berman M. Kinetic model for production and metabolism of very low density lipoprotein triglycerides. Evidence for a slow production pathway and results for normolipidemic subjects. J Clin Invest. 1979 Jun;63(6):1262-73. doi: 10.1172/JCI109421. PMID 221537
- [Result] Bjornson E, Packard CJ, Adiels M, Andersson L, Matikainen N, Soderlund S, Kahri J, Sihlbom C, Thorsell A, Zhou H, Taskinen MR, Boren J. Investigation of human apoB48 metabolism using a new, integrated non-steady-state model of apoB48 and apoB100 kinetics. J Intern Med. 2019 May;285(5):562-577. doi: 10.1111/joim.12877. Epub 2019 Mar 12. PMID 30779243
- [Derived] Taskinen MR, Matikainen N, Bjornson E, Soderlund S, Inkeri J, Hakkarainen A, Parviainen H, Sihlbom C, Thorsell A, Andersson L, Adiels M, Packard CJ, Boren J. Contribution of intestinal triglyceride-rich lipoproteins to residual atherosclerotic cardiovascular disease risk in individuals with type 2 diabetes on statin therapy. Diabetologia. 2023 Dec;66(12):2307-2319. doi: 10.1007/s00125-023-06008-0. Epub 2023 Sep 29. PMID 37775612

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After an initial telephone interview of 195 subjects, 77 were invited for a screening visit. Of these, 63 subjects were excluded because of failure to meet inclusion criteria.
Period: Overall Study
Arm/Group | Evolocumab
Started | 14
Completed | 13
Not Completed | 1
Not completed — worsening of asthma symptoms resulting in oral prednisolone use. | 1

BASELINE CHARACTERISTICS:
Population: Type II diabetic patients (a diagnosis of T2DM average duration 4.8 years). After an initial telephone interview of 195 subjects, 77 were invited for a screening visit. Of these, 63 subjects were excluded because of failure to meet inclusion criteria. All study subjects used daily stable doses of metformin and statin throughout the study period
Arm/Group | Evolocumab
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean ApoB Concentration Before and After Evolocumab
Description: Change in apolipoprotein B concentration in total plasma measured by using turbidimetric immunoassay.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
mg/dL
  Baseline | 75.9 (14.5)
  Week 12 | 35.3 (10.9)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Mean TRL-C Concentration Before and After Evolocumab
Description: Change in TRL-cholesterol concentration in plasma samples measured by using automated direct assay (Denka Seiken, Tokyo, Japan)
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
mg/dL
  Baseline | 33.4 (10.9)
  Week 12 | 17.8 (6.5)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Mean Total Production of ApoB48 Before and After Evolocumab
Description: Change in ApoB48 total production in plasma measured by using multicompartmental modeling. The power of mathematical modelling to describe the metabolic pathways of lipid and lipoprotein metabolism was demonstrated by Zech L et al (J Clin Invest 1979;63:1262-1273) and have been widely used over 30yrs. So far few studies have focused on the modelling of apo B48 and apo B100 after a meal that is more physiological than the fasting state (Björnson E et al. JIM 2019;285:562-577). Production rates for apo B48, apo B100 and triglycerides in chylomicrons, VLDL1 and VLDL2 were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90, 120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. Analysis of tracer/ tracee curves of stable isotopes was used to derived the estimates of kinetic parameters using a new mathematical modeling per day. These figures per day are used to report the data from this study.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: mg/d
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
mg/d
  Baseline | 570 (60)
  Week 12 | 580 (75)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.31, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Mean LDL FCR of ApoB100 Before and After Evolocumab
Description: Change in low-density lipoprotein fractional catabolic rate of ApoB100 in LDL from plasma samples measured by multicompartmental modeling. Production rates were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90, 120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. More detailed description see Outcome measure 3.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: pools/d
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
pools/d
  Baseline | 0.32 (0.15)
  Week 12 | 0.78 (0.34)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

5. Primary Outcome: LDL Pool Size of ApoB100 Before and After Evolocumab
Description: Change in low-density lipoprotein pool size of ApoB100 in LDL fraction prepared from plasma samples using density ultracentrifugation.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Evolocumab: Evolocumab 140 mg subcutaneous injection once every 2 weeks for 12 weeks
  Evolocumab
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
mg
  Baseline | 1500 (470)
  Week 12 | 460 (270)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Mean LDL-C Concentration Before and After Evolocumab
Description: Change in LDL-cholesterol concentration in plasma LDL fraction isolated by ultracentrifugation.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
mg
  Baseline | 1500 (470)
  Week 12 | 460 (270)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Mean ApoB48 Concentration Before and After Evolocumab
Description: Change in apolipoprotein B48 levels in total plasma measured by enzyme-linked immunosorbent assay.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
mg/L
  Baseline | 6.1 (3.8)
  Week 12 | 5.3 (3.3)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.27, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Mean CM TG-iAUC Before and After Evolocumab
Description: Change in chylomicron triglyceride incremental area under curve in plasma samples taken at particular time points after the meal. Area under the curve (AUC) was normalized so that 100% corresponds to the AUC before treatment; subsequently the percentage after treatment is in reference to this value. AUC values were calculated using the trapezoidal rule.
Time Frame: 0, 2, 4, 6, 8 hours after the meal at baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: (mmol/l)*h
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
(mmol/l)*h
  Baseline | 6.8 (3.6)
  Week 12 | 5.8 (4.4)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.22, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Mean ApoB48 AUC Before and After Evolocumab
Description: Change in apolipoprotein B48 area under curve in plasma samples taken at particular time points after the meal. Area under the curve (AUC) was normalized so that 100% corresponds to the AUC before treatment; subsequently the percentage after treatment is in reference to this value. AUC values were calculated using the trapezoidal rule.
Time Frame: 0, 2, 4, 6, 8 hours after the meal at baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: (mg/l)*h
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
(mg/l)*h
  Baseline | 66.8 (31.2)
  Week 12 | 57.4 (26.5)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.31, Kruskal-Wallis

10. Secondary Outcome: Mean VLDL1 ApoB100 Production Before and After Evolocumab
Description: Change in VLDL1 ApoB100 production rates measured from isolated VLDL from plasma samples using density ultracentrifugation and the enrichment of tracer was measured in isolated fractions following using mathematical modeling. Production rates were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90, 120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. More detailed description see Outcome measure 3.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: mg/d
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
mg/d
  Baseline | 790 (230)
  Week 12 | 750 (230)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.61, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Mean VLDL2 ApoB100 Production Before and After Evolocumab
Description: Change in VLDL2 apoB100 production rates measured from isolated VLDL2 from plasma samples by using density ultracentrifugation and the enrichment of tracer was measured in isolated fractions following using mathematical modeling. Production rates were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90, 120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. More detailed description see Outcome measure 3.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: mg/d
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
mg/d
  Baseline | 270 (91)
  Week 12 | 230 (96)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.11, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: IDL Pool Size of ApoB100 Before and After Evolocumab
Description: Change in intermediate-density lipoprotein pool size of ApoB100 in IDL fraction prepared from plasma samples using density ultracentrifugation.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
mg
  Baseline | 190 (50)
  Week 12 | 130 (49)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.003, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Mean IDL to LDL Transfer of ApoB100 Before and After Evolocumab
Description: Change in ApoB100 intermediate-density lipoprotein to low-density lipoprotein transfer in isolated samples from plasma by ultracentrifugation and measured using multicompartmental modeling. Production rates were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90, 120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. More detailed description see Outcome measure 3.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: mg/d
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
mg/d
  Baseline | 450 (190)
  Week 12 | 310 (140)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.027, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Mean VAT Before and After Evolocumab
Description: Change in visceral fat volume measured by magnetic resonance imaging
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: cm3
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
cm3
  Baseline | 2420 (960)
  Week 12 | 2450 (1100)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.84, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Mean Liver Fat Before and After Evolocumab
Description: Change in liver fat content measured by magnetic resonance imaging.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: fat %
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
fat %
  Baseline | 6.6 (6.6)
  Week 12 | 6.3 (7.2)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.59, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Mean SAT Before and After Evolocumab
Description: Change in subcutaneous fat volume measured by magnetic resonance imaging
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: cm3
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
cm3
  Baseline | 3900 (1700)
  Week 12 | 4110 (1600)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.81, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Mean VLDL1 Triglyceride Production Before and After Evolocumab
Description: Change in VLDL1 triglyceride production measured from isolated VLDL1 from plasma samples by using density gradient ultracentrifugation. Production rates were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90, 120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. More detailed description see Outcome measure 3.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: g/d
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
g/d
  Baseline | 34 (18)
  Week 12 | 33 (13)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.91, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Mean VLDL1 FCR of triglycerideBefore and After Evolocumab
Description: Change in VLDL1 fractional catabolic rate of triglyceride measured in isolated VLDL1 from plasma samples by using density ultracentrifugation and measured by multicompartmental modeling. Production rates were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90, 120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. More detailed description see Outcome measure 3.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: pools/d
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
pools/d
  Baseline | 38 (27)
  Week 12 | 37 (23)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 1, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Mean VLDL2 Triglyceride Total Production Before and After Evolocumab
Description: Change in VLDL2 triglyceride total production measured in isolated VLDL2 from plasma samples by using density ultracentrifugation and measured by multicompartmental modeling. Production rates were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90, 120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. More detailed description see Outcome measure 3.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: g/d
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
g/d
  Baseline | 8.8 (3.8)
  Week 12 | 8.5 (2.7)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.68, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Mean VLDL2 FCR of Triglyceride Before and After Evolocumab
Description: Change in VLDL2 fractional catabolic rate of triglyceride measured in isolated VLDL2 from plasma samples by using density ultracentrifugation and measured by multicompartmental modeling. Production rates were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90, 120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. More detailed description see Outcome measure 3.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: pools/d
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
pools/d
  Baseline | 10 (6.3)
  Week 12 | 15 (8.7)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.013, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Mean Postprandial CM of ApoB48 Before and After Evolocumab
Description: Change in Postprandial chylomicron of ApoB48 measured from plasma samples by liquid chromatography-mass spectrometry with multicompartmental modeling assay. Production rates were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90, 120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. More detailed description see Outcome measure 3.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: mg/d
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
mg/d
  Baseline | 240 (50)
  Week 12 | 230 (43)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.91, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Mean CM-apoB48 FCR of ApoB48 Metabolism Before and After Evolocumab
Description: Change in chylomicron-apoB48 fractional catabolic rate of ApoB48 in isolated chylomicrons from plasma samples measured by multicompartmental modeling assay. Production rates were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90, 120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. More detailed description see Outcome measure 3.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: pools/d
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
pools/d
  Baseline | 37 (24)
  Week 12 | 46 (32)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.27, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Mean CM-TG Production of ApoB48 Before and After Evolocumab
Description: Change in chylomicron-triglycerides production of ApoB48 in isolated chylomicrons from plasma samples measured by multicompartmental modeling assay. Production rates were derived from samples taken before and after the tracer injection and after the meal at 0, 30, 45, 60, 75, 90, 120, 150 min and at 3, 4, 5, 6, 8, 10, 24 hrs and averages for 24 hrs. More detailed description see Outcome measure 3.
Time Frame: Baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: g/d
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
g/d
  Baseline | 66.5 (0)
  Week 12 | 66.5 (0)

24. Secondary Outcome: Mean CM TG-AUC Before and After Evolocumab
Description: Change in chylomicron triglyceride area under curve in plasma at a particular time points after the meal. Area under the curve (AUC) was normalized so that 100% corresponds to the AUC before treatment; subsequently the percentage after treatment is in reference to this value. AUC values were calculated using the trapezoidal rule.
Time Frame: 0, 2, 4, 6, 8 hours after the meal at baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: (mmol/l)*h
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
(mmol/l)*h
  Baseline | 9.5 (4.9)
  Week 12 | 8.9 (5.9)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.84, Wilcoxon (Mann-Whitney)

25. Secondary Outcome: Mean ApoB48 iAUC Before and After Evolocumab
Description: Change in apolipoprotein B48 incremental area under curve in plasma at a particular time points after the meal. Area under the curve (AUC) was normalized so that 100% corresponds to the AUC before treatment; subsequently the percentage after treatment is in reference to this value. AUC values were calculated using the trapezoidal rule.
Time Frame: 0, 2, 4, 6, 8 hours after the meal at baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: (mg/l)*h
Arm/Group | Evolocumab
Number analyzed (Participants) | 13
(mg/l)*h
  Baseline | 18.4 (25.5)
  Week 12 | 13.9 (17.5)
Statistical Analysis 1: Comparison: Evolocumab; Test type: Other; p = 0.89, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: During 3 months of Evolocumab therapy
Groups:
- Evolocumab: Evolocumab 140 mg subcutaneous injection once every 2 weeks for 12 weeks
  Evolocumab: Evolocumab 140 mg subcutaneous injection once every 2 weeks for 12 weeks
Arm/Group | Evolocumab
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 3/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Evolocumab (N=13)
Blood glucose elevation (Blood and lymphatic system disorders) | 1 — No causality to Amgen drug used in this study
Non-cardiac chest pain (General disorders) | 1 — No causality to Amgen drug used in this study
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 — No causality to Amgen drug used in this study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Evolocumab (N=13)
Postural vertigo (Musculoskeletal and connective tissue disorders) | 1
Bradycardia (Cardiac disorders) | 1
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 9
Fungal nail disease (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Headache (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Skin eruption (Skin and subcutaneous tissue disorders) | 2
Hypertension (Blood and lymphatic system disorders) | 3
Bronchitis (Infections and infestations) | 1
Herpes simplex labialis (Infections and infestations) | 1
Tinnitus (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Tachycardia (Cardiac disorders) | 1
Pyuria (Renal and urinary disorders) | 1
Edema (Skin and subcutaneous tissue disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 2
Gastroenteritis (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Macrocytosis (Blood and lymphatic system disorders) | 1
Hematuria (Blood and lymphatic system disorders) | 1
Microcytosis (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT02948777/Prot_SAP_000.pdf